CLINICAL TRIAL: NCT02300714
Title: Fluoroscopically-guided Epidural Block in the Midthoracic Region: A Comparison of Anterioposterior Versus Oblique View Approach
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to lack of assistance and time to carry out the research.
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 4-2014-0822
Record Dates: First submitted 2014-11-20; First posted 2014-11-25 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Low Back Pain Requiring Epidural Injection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AP group (Active Comparator): oblique view approach during transforaminal epidural block
  Interventions: Procedure: oblique view approach
- OB group (Active Comparator): oblique view approach during transforaminal epidural block
  Interventions: Procedure: oblique view approach

INTERVENTIONS:
Procedure: oblique view approach

SUMMARY:
A comparison of anterioposterior versus oblique view approach method for fluoroscopically-guided epidural block in the midthoracic region. The investigators evaluate differences on total radiation time and technical feasibility between anterioposterior and oblique view approach method.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who were scheduled for the transforaminal epidural injection in midthoracic region (T5-T7)

Exclusion Criteria:

* Local anesthetic allergy, coagulopathy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-11; Primary Completion 2015-07-14 (Actual); Study Completion 2015-07-14 (Actual)

PRIMARY OUTCOMES:
Total radiation exposure time | immediately ≤1 sec after the confirmation of successful epidural injection
  Total radiation exposure time during whole epidural procedure.

SECONDARY OUTCOMES:
The number of the needle readjustments | immediately ≤1 sec after the confirmation of successful epidural injection
  The number of the needle readjustments for successful epidural injection

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, South Korea